CLINICAL TRIAL: NCT04738149
Title: A Proof of Concept, Split Study Measuring the Effectiveness of Topical ProstaglandinF2alpha, Microneedling and Excimer Laser in the Treatment of Vitiligo
Brief Title: Effect of Microneedling, Bimatoprost and Excimer in Vitiligo Treatment
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Principal Investigator, Joni Mazza Mccrann, Associate Professor, Medical University of South Carolina
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 00104695
Record Dates: First submitted 2021-01-22; First posted 2021-02-04 (Actual); Last update posted 2022-08-05 (Actual); Status verified 2022-08

CONDITIONS: Vitiligo
MeSH Terms: conditions — Vitiligo | interventions — Bimatoprost; Lasers, Excimer; Percutaneous Collagen Induction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Area 1: Excimer laser, bimatoprost, and microneedling (Experimental)
  Interventions: Drug: Bimatoprost; Device: Excimer laser; Device: Microneedling with a dermaroller
- Area 2: Excimer laser (Active Comparator)
  Interventions: Device: Excimer laser

INTERVENTIONS:
Drug: Bimatoprost — Participants will be receiving 2 drops per 4cm2 twice a week for 12 weeks
  Arms: Area 1: Excimer laser, bimatoprost, and microneedling
Device: Excimer laser — Participants will be receiving excimer laser 2x a week for 12 weeks
Device: Microneedling with a dermaroller — Participants will have 4cm2 area pre-treated with dermaroller 2x per week for 12 weeks
  Arms: Area 1: Excimer laser, bimatoprost, and microneedling

SUMMARY:
The purpose of this research is to treat vitiligo with a topical PGF2α, microneedling and excimer laser. The goal is to have greater repigmentation than the standard of care (excimer) after 12 weeks of treatment.

The study is a pilot, split study meaning the patient will receive one experimental and one standard of care treatment on symmetric lesions of similar location, geometrics and size.

Enrolled subjects will present biweekly to clinic on the same two days for twelve weeks. One lesion will be treated with microneedling, topical PGF2α and calibrated excimer laser, while the parallel lesion will be excimer laser alone. Physical exam, photographs, and a review of of the subjects medical records will occur in the study. Changes in size, appearance, and adverse events will be monitored throughout the study. The patient will also agree to close up photographs of their lesions throughout the study.

The possible benefit of joining this study is that the treatment received may be more effective than the other study treatment or then other available treatments for vitiligo, although this cannot be guaranteed.

ELIGIBILITY:
Inclusion Criteria:

* All patients 18 years and older with the diagnosis of Vitiligo.

Exclusion Criteria:

* Female patients currently pregnant or lactating
* Female patients with plans to come pregnant during the next 3 months
* Allergic reactions to topical or oral prostaglandins
* Uncontrolled skin disease
* History of glaucoma
* Concomitant disease or therapy that interferes with the diagnosis that might interfere with vitiligo diagnosis sand evaluation.
* Patients currently using other treatments for Vitiligo, such as topical steroids, calcineurin inhibitors, and Vitamin D analogs within 2 weeks of study initiation
* Inability or unwillingness of subject or legal guardian/representative to give

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2021-11-02 (Actual); Primary Completion 2022-05-15 (Actual); Study Completion 2022-05-15 (Actual)

PRIMARY OUTCOMES:
Percentage of skin repigmentation after 12 weeks | Post treatment (at week 12)
  A blinded outcome accessor will compare photographs of patients before and after treatment.
Number of patients with perceived improvement after 12 weeks. | Week 12
  Patients will be completing the Vitiligo Noticeability Scale that encompasses a series of questions assessing patient perceived change of before and after photographs.

SECONDARY OUTCOMES:
Change in quality of life | Baseline and post treatment approximately 12 weeks
  To access vitiligo patient specifically though a QOL reliable and valid scale.
Change in quality of life | Baseline and post treatment approximately 12 weeks
  To access quality of life via a validated general Dermatology Life Quality Index Scale.

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No